CLINICAL TRIAL: NCT06466746
Title: The Impact of Faba Bean Rich Bread on Iron Status, Postprandial Lipaemia and Satiety in Adults with Low Iron Stores
Brief Title: The Impact of Faba Bean Rich Bread on Iron Status, Postprandial Lipaemia and Satiety
Acronym: RtP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: King's College London (Other); University of Leeds (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor of Human Nutrition and Director of the Hugh Sinclair Unit of Human Nutrition, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UREC 24/02
Record Dates: First submitted 2024-06-04; First posted 2024-06-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anemia, Iron Deficiency; Cardiometabolic Disease; Low Iron Stores
Keywords: faba bean enriched bread; bioavailability; Enrichment of blood haemoglobin with Iron-57 stable isotope; Postprandial Lipaemia; Satiety; Visual analogue scales; Postprandial glycaemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Faba bean-enriched bread. (Active Comparator): 100 g of bread prepared using 40% faba bean flour and 60% wheat flour will be provided in the breakfast test meal.
  Interventions: Other: Raising the Pulse faba bean-enriched bread
- Conventional white bread (Placebo Comparator): 100 g of white bread prepared using 100% wheat flour will be provided in the breakfast test meal.
  Interventions: Other: Conventional White Bread

INTERVENTIONS:
Other: Raising the Pulse faba bean-enriched bread — 100 g of white bread produced using 40% faba bean enriched flour and 60% wheat flour will be provided in the breakfast meal with stork margarine, chocolate spread, a glass of orange juice and a glass of water containing the iron-57 stable isotope. An ad-libitum lunch consisting of pasta and a tomato sauce will be provide 6 hours after the breakfast.
  Arms: Faba bean-enriched bread.
Other: Conventional White Bread — 100 g of white bread produced using 100% wheat flour will be provided in the breakfast meal with stork margarine, chocolate spread, a glass of orange juice and a glass of water containing the iron-57 stable isotope. An ad-libitum lunch consisting of pasta and a tomato sauce will be provide 6 hours after the breakfast.
  Arms: Conventional white bread

SUMMARY:
High levels of animal proteins (meat) in the diet are linked with a greater risk of developing heart disease and other long-term health conditions. Recently there has been a shift to plant-based diets including plant proteins such as pulses, defined as beans, peas, chickpeas and lentils. Pulses are a nutritious and sustainable form of plant protein which are rich in fibre and iron. Despite this, the UK population does not consume the recommended daily amount of pulses (80g/day equivalent to a large handful). In contrast, bread is commonly consumed but very little is known about how bread enriched with pulses influences the amount of iron that is digested and absorbed by the body as well as risk factors for developing heart disease and type 2 diabetes.

The main purpose of this randomised controlled cross-over study is to determine how consuming bread enriched with pulses (in the form of faba bean flour at approximately 40% enrichment) compared with conventional white bread (100% wheat flour) influences the amount of iron absorbed in healthy males and females aged 18-50 years with low iron stores. Secondary aims are determining the effects on blood fats and sugar (glucose) and on feelings of fullness (also known as satiety) after eating the bread enriched in pulses and conventional white bread.

Participants will be required:

* To attend for seven study visits over a period of 60 days.
* Consume a breakfast meal containing either the faba bean-enriched bread or conventional bread over two study periods, each consisting of one 7 hour study visit and two consecutive visits of 2 hours in duration. After 28 days, participants will return for the second study period as above, with a final study visit conducted 28 days later.
* Give blood samples during 2 x 7 hour study visits
* Complete visual analogue scales to rate appetite after consuming the faba bean-enriched and conventional white bread.
* Record dietary intake prior to and during the study period.

DETAILED DESCRIPTION:
Since higher dietary intakes of animal protein (meat) are linked with heart disease and other long-term health problems, there has been a shift in recent years to consuming more plant-based foods. Legumes (e.g. beans) provide a sustainable and nutritious source of protein and are higher in fibre and micronutrients (such as iron) compared with staple cereals. Higher intakes of pulses lower blood sugar and fat levels, increase feelings of fullness (satiety) and reduce blood pressure. The higher iron content in mature faba beans may also help to reduce iron-deficiency anaemia, the most common diet-related deficiency. However, studies have suggested that the absorption of iron from pulses (known as bioavailability) is lower than from meat due to the presence of compounds in plants that interfere with absorption (anti-nutrients). Processing techniques such as milling of faba beans are considered to lower or even eliminate these compounds. In the Raising the Pulse (RtP) project, flour milled from homegrown faba beans will be used to produce a pulse-enriched loaf which could be adopted in the UK diet and benefit both health and the environment. However, very little is known about how bread enriched with pulses may influence firstly, iron bioavailability and secondly, blood sugar and fat levels which are common risk factors for developing heart disease and diabetes.

This randomised controlled cross-over study will aim to recruit 16 healthy, non-anaemic males and females with low iron stores. Aside from the screening visit where participants will be assessed for eligibility and consent for participation gained, this study will involve seven study visits. The first study visit (Day 1) will be approximately 7 hours (420 minutes) in duration and participants will be randomly assigned to consume either the faba bean-enriched bread or the conventional white bread along with a drink containing iron-57, a naturally occurring non-radioactive form of iron found in very low levels in the diet (stable isotope) to measure iron absorption. Blood samples will be collected to measure blood haemoglobin, sugar and fat levels as well as hormones known to impact appetite, and participants will be asked to complete visual analogue scales to rate their appetite. At the visit, an ad-libitum (unrestricted) meal will be provided 6 hours after eating the test breakfast and the amount of food eaten will be used to assess satiety. Participants will then return on days 2 and 3 to consume the same test meal and complete visual analogue scales to rate appetite for 2 hours. At day 30, participants will return for the second 7 hour (420 minute) study visit to consume the other type of bread and return on days 31 and 32 for the shorter study visits. The day 30 fasting blood sample will be used to measure the enrichment of blood haemoglobin with iron-57 to determine the amount of iron absorbed from the test bread given on day 0. On day 60, participants will return to the clinical unit to give a final fasting blood sample to measure iron bioavailability (enrichment of blood haemoglobin with iron-57) from the test bread given on day 30. Dietary intake will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Non-anaemic, males and pre-menopausal females (must have regular periods)
* Aged 18-50 years old
* BMI between 19 - 30 kg/m2
* Low iron stores (serum ferritin between 13-40 µg/L for females and 30-90 µg/L for males)

Exclusion Criteria:

* Food allergies or intolerances to faba beans (favism) or gluten
* Diagnosed with anaemia (haemoglobin <115 g/L for females or <130 g/L for males) or haemochromatosis
* C-reactive protein (>3mg/L)
* Smokers
* A history of alcohol abuse (> 14 units/ week)
* CVD or medical history of MI or stroke in the past 12 months
* Diabetes (fasting glucose >7.0 mmol/L)
* Kidney, liver, pancreas or intestinal disease, gastrointestinal disorder or use of drugs likely to alter gastrointestinal function
* Pregnancy, planning a pregnancy in the next six months or breastfeeding
* Peri- and post-menopausal women or women with irregular periods
* Planning on a weight-reducing regimen (lost >3kg in last 6 months)
* Parallel participation in another intervention study
* Hypertension (blood pressure > 140/90 mmHg), cancer, taking medication for hyperlipidaemia (statins), or inflammation
* Taking vitamin or mineral supplements
* Donated blood in the last 3 months
* Any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention and metabolic study (such as a pacemaker)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the enrichment of whole blood haemoglobin with iron-57 stable isotope 30 days after consuming the faba bean-enriched bread and conventional bread. | Day 0 (baseline), day 30 and day 60
  The measurement of iron-57 in whole blood is a validated method for determining the absorption of iron from the bread given in the test meals (also known as bioavailability)

SECONDARY OUTCOMES:
Fasting concentrations of iron status markers | Day 0 (baseline), day 30 and day 60
  Serum ferritin (a measure of the level of iron stored by the body) and soluble transferrin receptor (a measure of functional iron status) will be measured by immunoassay.
Fasting concentration of C-reactive protein (a marker of inflammation) | Day 0 (baseline), day 30 and day 60
  Inflammation, which is characterised by the acute-phase response to infection, can directly affect the concentrations of most iron status markers. C-reactive protein will be measured in the fasting blood sample collected at each study visit to aid the interpretation of the data for the iron status markers.
Fasting levels of the full blood count parameters | Day 0 (baseline), day 30 and day 60
  The level of white blood cells, red blood cells, platelets, haematocrit and haemoglobin in the whole blood sample will be measured using a haematology analyser.
Fasting concentration of total cholesterol, high-density lipoprotein-cholesterol, triacylglycerol and non-esterified fatty acids. | Day 0 (baseline), day 30 and day 60
  Serum lipids will be measured directly using a clinical chemistry analyser.
Fasting low-density lipoprotein-cholesterol concentration | Day 0 (baseline), day 30 and day 60
  The low-density lipoprotein-cholesterol concentration will be calculated from the total cholesterol, high-density lipoprotein-cholesterol and triacylglycerol concentrations using the Friedewald formula.
Postprandial concentrations of lipids after consuming the faba bean-enriched bread and control bread. | Acute study on Days 0 and 30, blood taken prior to eating the test meal (0 minutes) and then at 15, 30, 45, 60, 90, 120, 180, 240, 300 and 360 minutes post meal ingestion.
  Serum triacylglycerol and non-esterified fatty acids will be measured in the postprandial blood samples collected for 360 minutes after each acute test meal.
Fasting glucose concentration | Day 0 (baseline), day 30 and day 60
  Serum glucose will be measured using a clinical chemistry analyser.
Fasting insulin concentration | Day 0 (baseline), day 30 and day 60
  Serum insulin will be measured using an enzyme-lined immunosorbent assay.
Fasting estimate of insulin resistance | Day 0 (baseline), day 30 and day 60
  HOMA-IR (Homeostasis model assessment estimated insulin resistance) will be calculated using the glucose and insulin data.
Fasting estimate of insulin sensitivity | Day 0 (baseline), day 30 and day 60
  QUICKI (Quantitative Insulin Sensitivity Check Index) will be calculated using the glucose and insulin data.
Postprandial glucose concentrations after consuming the faba bean-enriched bread and control bread. | Acute study on Days 0 and 30, blood taken prior to eating the test meal (0 minutes) and then at 15, 30, 45, 60, 90, 120, 180, 240, 300 and 360 minutes post meal ingestion
  Serum glucose will be measured in the postprandial blood samples collected for 360 minutes after each acute test meal.
Postprandial insulin concentrations after consuming the faba bean-enriched bread and control bread. | Acute study on Days 0 and 30, blood taken prior to eating the test meal (0 minutes) and then at 15, 30, 45, 60, 90, 120, 180, 240, 300 and 360 minutes post meal ingestion
  Serum insulin will be measured in the postprandial blood samples collected for 360 minutes after each acute test meal.
Fasting and postprandial concentrations of gut hormones | Acute study on Days 0 and 30, blood taken before meal ingestion at 0 minutes and then at 15, 30, 45, 60, 90, 120, 180, 240, 300 and 360 minutes post meal ingestion
  C-peptide, PYY, GIP and GLP-1 will be measured using a Luminex multiplex assay.
Fasting apolipoprotein B concentration | Day 0 (baseline), day 30 and day 60
  Serum apolipoprotein B will be measured using a clinical chemistry analyser.
Postprandial apolipoprotein B concentrations after consuming the faba bean-enriched bread and control bread. | Acute study on Days 0 and 30, blood taken prior to eating the test meal (0 minutes) and then at 60, 120, 180, 240, 300 and 360 minutes post meal ingestion.
  Serum apolipoprotein B concentrations will be measured using a clinical chemistry analyser.
Fasting and postprandial concentrations of amino acids | Acute study on Days 0 and 30, blood taken before eating the test meal (0 minutes) and then at 15, 30, 45, 60, 90, 120, 180, 240, 300 and 360 minutes post meal ingestion
  Individual amino acids
Height | Day 0 (baseline)
  Height will be measured to the nearest cm using a stadiometer
Body weight | Day 0 (baseline), day 30 and day 60
  Body weight will be measured using a Tanita scale.
Body fat percentage | Day 0 (baseline), day 30 and day 60
  Body fat percentage will be measured using a Tanita scale by bioelectrical impedance.
Body fat mass and lean mass | Day 0 (baseline), day 30 and day 60
  Body fat mass and lean mass will be measured using a Tanita scale by bioelectrical impedance.
Body mass index calculation | Day 0 (baseline), day 30 and day 60
  Body mass index will be calculated using the body weight (kg) and height data (m).
Waist and hip circumferences | Day 0 (baseline), day 30 and day 60
  A non-stretch tape measure will be used to measure the waist and hip circumferences in cm.
Clinic blood pressure | Day 0 (baseline), day 30 and day 60
  Systolic blood pressure, diastolic blood pressure and pulse pressure
Postprandial feelings of satiety_7 hour study visit (long day) | Acute study on Days 0 and 30, prior to eating the test meal (0 minutes) and then at 15, 30, 60, 120, 240 and 360 minutes post meal ingestion
  100 mm visual analogue scale. This scale is well validated for measuring appetite and satiety. Each rating score is out of 100.
Postprandial feelings of satiety_2 hour study visit (short day) | Days 1, 2, 31 and 32 prior to eating the test meal (0 minutes) and then at 15, 30, 60 and 120 minutes post meal ingestion.
  100 mm visual analogue scale. This scale is well validated for measuring appetite and satiety. Each rating score is out of 100.
Habitual dietary intake of the study participants | Day 0 (baseline), day 30 and day 60
  Record of food and drink intake prior to each study visit.
Fasting blood samples stored for future ethically approved research related to the project aims and objectives. | Day 0 (baseline), day 30 and day 60
  Spare whole blood and plasma/serum samples will be collected and biobanked for future research
Postprandial blood samples stored for future ethically approved research related to the study aims and objectives. | Acute study on Days 0 and 30, blood taken prior to eating the test meal (0 minutes) and then at 15, 30, 45, 60, 90, 120, 180, 240, 300 and 360 minutes post meal ingestion.
  Spare plasma/serum samples will be biobanked for future research

CONTACTS AND LOCATIONS:
Overall Officials: Abbe Davy, BSc, Study Director — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All anonymised IPD that underlie results in a publication and analytic code for the statistical analysis.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Anonymised data will be made available on reasonable request one year after manuscripts have been published.
Access Criteria: For data sharing and preservation, anonymised IPD will be archived in the University of Reading Research Data Archive. Access will be overseen by the project PI. This information will be maintained under Professor Julie Lovegrove's and Dr Kim Jackson's authority and disposed of appropriately by the PI [Professor Julie Lovegrove]. If the PI should leave the University, the Personal Information will be under the authority of the Head of School.

REFERENCES:
- [Background] Lovegrove JA, O'Sullivan DM, Tosi P, Millan E, Todman LC, Bishop J, Chatzifragkou A, Clegg ME, Hammond J, Jackson KG, Jones PJ, Lignou S, Macready AL, McMeel Y, Parker J, Rodriguez-Garcia J, Sharp P, Shaw LJ, Smith LG, Tebbit M. 'Raising the Pulse': The environmental, nutritional and health benefits of pulse-enhanced foods. Nutr Bull. 2023 Mar;48(1):134-143. doi: 10.1111/nbu.12601. Epub 2023 Jan 17. PMID 36649740